CLINICAL TRIAL: NCT02582359
Title: Phase I Dose Escalation Study of Millennium 9708 in Combination With Induction and Consolidation Chemotherapy in Adults >= 60 Years With Acute Myeloid Leukemia
Brief Title: MLN 9708 in Induction and Consolidation for Adults With AML >= 60 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Philip C. Amrein, M.D., Philip C. Amrein, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-276
Record Dates: First submitted 2015-10-18; First posted 2015-10-21 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ixazomib; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MLN9708 (Experimental): Phase I dose escalation study of MLN9708 with induction chemotherapy
  * MLN9708 -oral on predetermined days per cycle
  * Cytarabine, continuous infusion for predetermined duration and dosage
  * Daunorubicin short IV infusion or rapid injection for predetermined
  Phase I dose escalation study of MLN9708 with consolidation chemotherapy after establishment of MTD with induction
  Interventions: Drug: MLN9708; Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: MLN9708 — Dose of 1.5 mg or 2.3 mg or 3.0 mg taken by mouth on days 2, 5, 9, 12 of each cycle.
  Other Names: Ixazomib
Drug: Cytarabine — Induction: cytarabine 100 mg/m2/day continuous infusion, days 1-7 Consolidation: cytarabine 2000 mg/m2/day, 3 hour infusion, on days 1-5
  Other Names: Cytosar-U®; Ara-C; Arabinosylcytosine
Drug: Daunorubicin — Daunorubicin 60 mg/m2, IV bolus, on days 1-3 of induction, only.
  Other Names: Cerubidine®

SUMMARY:
This research study is evaluating drugs called Millennium 9708 (referred to as MLN9708) in combination with standard therapy for acute myeloid leukemia (AML) consisting of daunorubicin and cytarabine as a possible treatment for the patient AML.

DETAILED DESCRIPTION:
This research study is a clinical trial comprised of two Phase I portions an induction treatment (initial treatment), and a consolidation treatment (which is given later). The patient is being asked to participate in one or both phase I portions of this study.

A phase I study tests the safety of an investigational drug or combination of drugs. Phase I studies also try to define the appropriate dose of the investigational drugs to use for further studies. "Investigational" means that the drug combination is being studied. It also means that the FDA (U.S. Food and Drug Administration) has not approved the drug combination for the participant's type of cancer.

In this research study, the investigators are studying the safety and tolerability of MLN9708 in combination with standard treatment for adults 60 years of age or older with AML.

In the first phase I portion of treatment ("induction") participants will receive MLN9708 in combination with daunorubicin and cytarabine. Once the maximally tolerated dose (MTD) of MLN9708 is established in this induction portion, up to 36 additional participants will be enrolled in the portion focusing on consolidation.

The drugs daunorubicin and cytarabine have been approved by the FDA (U.S. Food and Drug Administration). MLN9708 is not approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 60 years or older.
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.]
* Patients must have a diagnosis of AML according to the World Health Organization (WHO) criteria. Therapy-related and secondary AML (arising after a period of myelodysplasia [MDS]) allowed. Prior treatment for MDS with hypomethylator-based therapy and lenalidomide allowed, but not allowed if used after the diagnosis of AML is made, since enrollment to this study is not for relapsed AML.
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2. Performance status of 3 permissible if related to disease.
* Patients must meet the following clinical laboratory criteria:

  * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN) unless related to disease or patient known to have underlying Gilbert's disease.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 ULN.
  * Calculated creatinine clearance ≥ 30 mL/min (see Section 12.2).

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Failure to have fully recovered (ie, ≤Grade 1 toxicity) from the reversible effects of prior chemotherapy as stated in Section 5.1.4.
* Major surgery within 14 days before enrollment.
* Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708.
* Suspected AML-related central nervous system involvement. A lumbar puncture (LP) is not required to exclude central nervous system (CNS) disease.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has ≥ Grade 1 neuropathy, sensory, with or without pain, motor, or autonomic, on clinical examination during the screening period.
* Participation in other clinical trials involving investigational agents within 21 days of the start of this trial and throughout the duration of this trial.
* Prior chemotherapy treatment for AML (Prior treatment with hydroxyurea and/or leukapheresis to control white blood cell count acceptable). Prior chemotherapy for MDS or myeloproliferative neoplasms (MPN) such as azacitidine, decitabine, and thalidomide, is permitted, but such treatments once MDS or MPN has transformed to AML is not permitted.
* Acute promyelocytic leukemia(APL) by WHO criteria [AML with t(15;17)]
* Cardiac ejection fraction (EF) < 40%
* Systemic treatment, during or within 48 hours of the first dose of MLN9708, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort. The washout period will be extended to 2 days if patients are receiving extended release ciprofloxacin. For this protocol prophylactic antibiotics are not recommended, at least not until 48 hours after the last dose of study drug (given on Day 12), when the patient may be neutropenic. For patients with fever and/or infections, cefepime and ambisome are acceptable.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
MTD/recommended phase 2 dose (RP2D) of MLN9708 in combination with induction chemotherapy | 1 year
  Safety of MLN9708 in induction
MTD/RP2D of MLN9708 with combination with consolidation chemotherapy | 1 year
  Safety of MLN9708 in consolidation tested separately

SECONDARY OUTCOMES:
Dose Limiting Toxicities of MLN9708 | 1 year
  Generally by NCI CTCAE: grade 3 neuropathy, grade 3 non-hematological toxicity that does not resolve to grade 2, grade 4 hematological toxicity not due to persistent AML that persists
Disease Free Survival (DFS) | 2 Years: Complete remission (CR) or complete remission without platelet recovery (CRp) to relapse or death, whichever comes first, for patients who receive study drug in induction and regardless of consolidation therapy
  Duration in weeks or months from determination of remission to time of relapse or death
Overall Survival (OS) | 2 Years
  Duration in weeks or months from day 1 of protocol treatment to time of death
Remission Rate | 2 years
  Percentage of patients starting day 1 treatment that achieve a remission (CR or CRp)
Relationship between CD74 expression and remission, DFS, OS | 2 Years
  Degree of CD74 expression on leukemia blasts compared to the rate of remission and length of DFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Amrein, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States